CLINICAL TRIAL: NCT03326960
Title: Effects of Anesthetics Sevoflurane, Propofol and Desflurane on Postoperative Delirium (POD) and Postoperative Cognitive Disorder (POCD)
Brief Title: Sevoflurane, Propofol and Desflurane on POD/POCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Head of Psychiatry, Shanghai 10th People's Hospital
Other Study IDs: dsyy002
Record Dates: First submitted 2017-10-06; First posted 2017-10-31 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Sevoflurane; Propofol; Desflurane
Keywords: general anesthesia; postoperative delirium; postoperative cognitive dysfunction; retinal nerve fiber layer; biomarker
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Sevoflurane; Propofol; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will collect 10ml venous blood before anesthesia, and then 10ml venous blood after surgery on Day 1, Day 2 and Day 3, respectively. Serum level of vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) will be tested.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sevoflurane: Patients in Sevoflurane group are maintained with sevoflurane from an anesthesia machine through the laryngeal mask airway guided by Narcrotrend index monitoring.
  Interventions: Drug: Sevoflurane
- Propofol: Patients in Propofol group are maintained with propofol through intravenous administration guided by Narcrotrend index monitoring.
  Interventions: Drug: Propofol
- Desflurane: Patients in Desflurane group are maintained with desflurane from an anesthesia machine through the laryngeal mask airway guided by Narcrotrend index monitoring.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia maintenance with sevoflurane guided by Narcrotrend index monitoring.
  Groups: Sevoflurane
Drug: Propofol — Anesthesia maintenance with propofol guided by Narcrotrend index monitoring.
  Groups: Propofol
Drug: Desflurane — Anesthesia maintenance with desflurane guided by Narcrotrend index monitoring.
  Groups: Desflurane

SUMMARY:
The investigators will perform clinical studies to test the hypothesis that participants who have total hip/knee replacement under sevoflurane, propofol or desflurane anesthesia will have different effects on the incidence and severity of POD/POCD, and POD/POCD is associated with retinal nerve fiber layer (RNFL) thickness, as well as Serum level of vitamin B12, folic acid, homocysteine and human myeloid differentiation protein-2 (MD-2s). The investigators plan to perform the studies in 300 participants at Shanghai 10th People's Hospital.

DETAILED DESCRIPTION:
Postoperative delirium (POD) and postoperative cognitive disorder (POCD) are the most common complications of geriatric surgical patients, which could cause long-term social dysfunction, high mortality and increased medical cost. Currently, there is no efficient biomarker for POD/POCD, and it also remains largely unknown whether different anesthesia might lead to different incidence and severity of POD/POCD. The investigator's previous studies showed that thickness of retinal nerve fiber layer thickness (RNFL-T) measured by optical coherence tomography (OCT) was associated with POD/POCD; change of RNFL thickness (RNFL-C) in certain period correlated with cognitive deterioration. Thus, the investigators consider that RNFL might be a potential biomarker of POD/POCD. In the proposed large-scale longitudinal studies, the investigators will clinically validate RNF-LT as pre-operative POD/POCD biomarker, and RNFL-C as post-operative biomarker of POD/POCD. Finally, the investigators will compare the effects of surgery (total hip/knee replacement) under general anesthesia with sevoflurane, propofol and desflurane on the incidence and severity of POD/POCD in patients. Results from the proposed studies will likely establish RNFL as a potential POD/POCD biomarker, promote the clinical utilization of OCT-RNFL in early screening and outcome prediction of POD/POCD, and finally optimize anesthesia care of geriatric surgical patients to avoid or reduce POD/POCD incidence. These findings will lead to better postoperative outcomes of geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or older
* Chinese Mandarin as the native language
* scheduled to undergo hip/knee surgery under general anesthesia
* American Society of Anesthesiologists (ASA) class I-Ⅲ

Exclusion Criteria:

* Prior diagnoses of neurological diseases according to ICD-10
* History of severe psychiatric disorders according to DSM-IV
* Visual or auditory defects
* Participating in the investigation of another study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged 60 years old or older, who admitted to the Department of Orthopedics at Shanghai 10th People's Hospital and had been scheduled to undergo knee or hip fractures were screened and asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | At 1st day after the surgery
  Postoperative delirium will be determined by Confusion Assessment Method (CAM) at 1st postoperative day

SECONDARY OUTCOMES:
Postoperative delirium | At 2nd day after the surgery
  Postoperative delirium will be determined by CAM at 2nd postoperative day
Postoperative delirium | At 3rd day after the surgery
  Postoperative delirium will be determined by CAM at 3rd postoperative day
Preoperative cognitive function | Preoperative cognitive function (baseline)
  Preoperative cognitive function will be assessed by neuropsychological battery
Postoperative cognitive dysfunction | Change from baseline cognitive dysfunction at 1 week
  Postoperative cognitive dysfunction will be assessed by neuropsychological battery before and after the surgery and anesthesia
Postoperative cognitive dysfunction | Change from baseline cognitive dysfunction at 3rd month
  Postoperative cognitive dysfunction will be assessed by neuropsychological battery
Retinal nerve fiber layer thickness | Change from baseline RNFL thickness at 3rd month
  Retinal nerve fiberlayer（RNFL）thickness will be measured by optical coherence tomography (OCT) before and after surgery and anesthesia
Serum level of vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) | Before the surgery (baseline)
  vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) will be tested
Serum level of vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) | At 1st day after the surgery
  vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) will be tested
Serum level of vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) | At 2nd day after the surgery
  vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) will be tested
Serum level of vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) | At 3rd day after the surgery
  vitamin B12, folic acid, homocysteine and myeloid differentiation protein-2 (MD-2s) will be tested

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, M.D.,Ph.D, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vlisides P, Xie Z. Neurotoxicity of general anesthetics: an update. Curr Pharm Des. 2012;18(38):6232-40. doi: 10.2174/138161212803832344. PMID 22762477
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Gleason LJ, Schmitt EM, Kosar CM, Tabloski P, Saczynski JS, Robinson T, Cooper Z, Rogers SO Jr, Jones RN, Marcantonio ER, Inouye SK. Effect of Delirium and Other Major Complications on Outcomes After Elective Surgery in Older Adults. JAMA Surg. 2015 Dec;150(12):1134-40. doi: 10.1001/jamasurg.2015.2606. PMID 26352694
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092